CLINICAL TRIAL: NCT01229709
Title: Phase 2 Mindfulness Based Tinnitus Reduction (MBTR) Study: A Symptom Perception Shift Program
Brief Title: Mindfulness Based Tinnitus Reduction (MBTR): A Symptom Perception Shift Program
Acronym: MBTR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8935-35834-01
Record Dates: First submitted 2010-10-26; First posted 2010-10-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Tinnitus; Anxiety; Depression
Keywords: Tinnitus; Mindfulness; MBSR; Mindfulness Based Stress Reduction; MBTR
MeSH Terms: conditions — Tinnitus; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness Based Tinnitus Reduction (Experimental)
  Interventions: Behavioral: Mindfulness Based Tinnitus Reduction
- Tinnitus Counseling Only Control (No Intervention): Control group subjects will have had treatment as usual (TAU) care from the UCSF Audiology Clinic which includes Tinnitus Counseling (TC) at least three-months prior to enty into the study.

INTERVENTIONS:
Behavioral: Mindfulness Based Tinnitus Reduction — The Mindfulness Based Tinnitus Reduction (MBTR) program will be held for two-and-a-half hours one evening per week over 8 consecutive weeks. Participants will also complete a day-long Sunday retreat between the 6th and 7th sessions. Each participant will take part in a 30-minute private interview with the course instructor prior to beginning the program.
  Other Names: MBTR
  Arms: Mindfulness Based Tinnitus Reduction

SUMMARY:
This study is a randomized, controlled trial of Mindfulness Based Tinnitus Reduction (MBTR) vs. Treatment As Usual (TAU). This study aims to determine patient's benefit from participating in an 8-week MBTR program as measured by a reduction in clinical symptoms, if present, and a tinnitus symptom perception shift. Sixty-four tinnitus patients who have previously received Tinnitus Counseling (TAU) at the UCSF Audiology Clinic under the direction of Robert Sweetow, PhD will be invited to participate in the MBTR study. Subjects will be randomly assigned to the experimental and control groups of 32 each. All subjects will have received Tinnitus Counseling at least 6-months prior to entry into the study. Tinnitus symptom activity and discomfort as well as psychological outcomes will be assessed by self-report questionnaires. The primary outcome measure is the Tinnitus Handicap Inventory (THI) measuring tinnitus symptom severity. The secondary outcome measures include the Tinnitus Visual Analogue Scale (TVAS), the Symptom Checklist-90-Revised (SCL-90-R), Hamilton Anxiety and Depression Scale (HADS), and the Five Factor Mindfulness Questionnaire (FFMQ). In addition to tinnitus symptom severity, secondary outcome measures are used to measure change in mindfulness and other clinical symptoms such as anxiety and depression, if they exist. The experimental group will complete measures at pre-, post-, at 3-months and 12-months follow-up. A 12-month follow-up assessment will be conducted with the experimental group to identify any enduring effects of the treatment. The control group will fill out measures at pre-, post-, and 3-month time periods. The 12-month follow-up will be conducted with the experimental group only and will be the uncontrolled portion of the study.

The purpose of this study is to 1) Design and execute an MBTR program for patients with tinnitus within the UCSF Department of Audiology. 2) Determine patient's benefit from participating in an 8-week MBTR program as measured by a decrease in tinnitus distress, and a reduction in clinical symptoms (i.e., depression, anxiety), if present. 3) Compare the responses on study measures to those of the control group. 4) Collect follow-up data at 6- and 12-months post intervention to assess enduring effects, if any, in the experimental group. 5) Use the data and patient feedback to modify UCSF's Audiology program and guide future programming in regards to the treatment and care of patients with tinnitus.

DETAILED DESCRIPTION:
Tinnitus is a medical term for acoustical perceptions heard in the ear(s) or head, not produced by external sound. This sound can be experienced as a ringing, buzzing, whooshing, or hissing. Estimates suggest that as many as 50 million people in the United States experience tinnitus to some degree. Approximately 12 million of these people experience tinnitus bothersome enough to seek medical treatment. Two to 3 million Americans are severely affected by their tinnitus to the extent that their ability to function is severely impaired.

Mindfulness Based Stress Reduction (MBSR) is an established treatment with broad applicability to clinical science. MBSR has been scientifically shown to improve well-being and health in the treatment of depression (Mason O, Hargreaves I. 2001), anxiety (Kabat-Zinn, et al 1992), stress (Kabat-Zinn, et al. 1992), fibromyalgia (Grossman, et al. 2007), chronic fatigue (Surawy, et al. 2005), psoriasis (Kabat-Zinn, et al. 2003), treatment of cancer (Speca, et al. 2006), multiple schlerosis (Grossman, et al. 2010), and pain (Kabat-Zinn, et al. 1985).

Treatments used for pain management are of particular interest to those studying tinnitus because many similarities between individuals suffering with tinnitus and pain can be drawn. Both pain and tinnitus patients commonly express a perceived lack of control over their symptoms, problems with aspects of attention and focus, maladaptive coping strategies, catastrophic thinking, and the use of similar treatment methods (e.g., cognitive coping strategies, CBT, relaxation techniques)(Moller, 2000, Tonndorf, 1987). Like intractable pain, there is no single identifiable cause of tinnitus, there is no single medical or surgical treatment that is effective, there are a wide range of psychological effects, and one's lifestyle and general health are particularly affected. One of the first studies looking at mindfulness as a means of pain management was conducted by Jon Kabat-Zinn, Lipworth, and Burney (1985). They took 90 patients with chronic pain and trained them in a ten-week stress reduction and relaxation program. Significant reductions in present moment pain, negative body image, inhibition of activity by pain, mood disturbance such as anxiety and depression were shown. Significant improvements in activity level and feelings of self-esteem were also reported. Reductions and improvements were maintained 15-months post-treatment. Due to the success of mindfulness-based interventions with chronic pain, the healing benefits of mindfulness are being translated to tinnitus care in this study.

To date only one pilot study has been conducted using mindfulness meditation as a treatment for tinnitus. A study conducted in Wales by Sadlier, Stephens, & Kennedy (2008) used a combination of cognitive behavioral therapy and mindfulness meditation to treat 25 individuals with chronic tinnitus. The subjects were split into two groups. The treatment group received four one-hour sessions of CBT and Mindfulness Meditation practice while the second group waited 3-months and was then treated with the same intervention. Significant reductions in tinnitus post-treatment and at 4 to 6 months follow-up were recorded. The proposed MBTR study isolates mindfulness from CBT approaches to tinnitus, and may be an important contribution to the clinical literature on the care of tinnitus.

Introduction and Specific Aims This study aims to determine the efficacy of MBTR in reducing symptoms of tinnitus in adults. Primary objectives include: 1) Design and execute an MBTR program within the UCSF Department of Audiology for patients with tinnitus. 2) Determine patient's benefit from participating in an 8-week MBTR program as measured by a reduction in clinical symptoms, if present, and a tinnitus symptom perception shift. 3) Compare the responses on study measures to those of the control group. 4) Use the data and patient feedback to modify UCSF's Audiology program and guide future programming in regards to the treatment and care of patients with tinnitus.

The above mentioned objectives will be met through testing the following primary hypotheses:

Hypothesis 1a: MBTR + TAU will be more effective than TAU alone in reducing tinnitus symptoms (25-item Tinnitus Handicap Inventory [THI]) in adult patients with chronic tinnitus over an 8-week period.

Hypothesis 1b: MBTR + TAU will be more effective than TAU alone in reducing tinnitus symptoms (25-item Tinnitus Handicap Inventory [THI]) in adult patients with chronic tinnitus at 3-months follow-up.

Hypothesis 1c: Reduction in tinnitus symptoms (25-item Tinnitus Handicap Inventory [THI]) in the MBTR + TAU will be maintained at 12-months follow-up.

Secondary hypotheses and analyses are as follows:

Hypothesis 2: Effect on Functional Status: MBTR + TAU will be more effective than TAU alone in reducing anxiety and depressive symptoms, if they exist (17-item Hamilton Anxiety and Depression Scale [HADS]) and in reducing additional clinical symptoms, if they exist (90-item Symptom Checklist-90-Revised [SCL-90-R]) and enhanced mindfulness (39-item Five Factor Mindfulness Questionnaire [FFMQ]).

Hypothesis 3: Mediators of MBTR Efficacy: The effect of MBTR on tinnitus severity (THI, Tinnitus Visual Analogue Scale [TVAS]) and functional status (HADS and SCL-90-R) will be mediated by enhanced mindfulness (FFMQ).

Hypothesis 4: Length of Efficacy: We will assess whether treatment gains in tinnitus severity (THI, TVAS), functional status (HADS, SCL-90-R), and mindfulness (FFMQ) are retained at 3-months and at 12-months follow-up for the experimental group.

Research Design and Methods Subject Recruitment A chart review of past patients (approximately 700) from the UCSF Audiology Clinic who have been seen for Tinnitus Counseling (Treatment as Usual-TAU) at least six-months prior to enrollment in the study will take place. A list of the inclusion/exclusion criteria are below.

Inclusion Criteria

Subject Characteristics

* Age > 18
* English speaking
* Duration of subjective chronic tinnitus > 6 months
* Received Tinnitus Counseling (TAU) at the UCSF Audiology Clinic > 6 months prior to entering the study
* Moderate to strong tinnitus annoyance (Minimum THI score of > 24 per chart review)

Exclusion Criteria

Subject Characteristics

* Age < 18
* Non-English speaking
* > Moderate Hearing Loss
* Duration of chronic subjective tinnitus < 6 months
* Severe depression and/or anxiety (as measured by the HADS)
* Recent (within 3-month) history of alcohol or drug abuse or dependence other than tobacco or caffeine
* No recent (within 3 months) start of new tinnitus treatment
* History of psychotic disorders or dementia
* THI score < 24
* Currently undergoing litigation or legal matters related to auditory disorders

Three hundred letters will be mailed to those patients from the Clinic's database who meet inclusion criteria and have been seen for tinnitus counseling at least six-months prior to entry into the study. Patients will respond via postcard as to whether they would like to learn more about the study. Patients will be informed in the letter that if no response is received via postcard to the Clinic within two weeks, a research assistant will follow up with a phone call as a reminder to respond. To prevent over-enrollment/recruitment of subjects, letters will be sent out in waves of 100 at a time. Recruitment will stop when 80 patients respond to participate (a 20% drop out-rate is expected bringing the number down to 64).

The 80 patients who express interest in participating in the study and meet inclusion criteria per chart review will be invited to take part in a 30-minute individual interview with one of the two MBTR course instructors prior to beginning the program. The 30-minute individual interview will serve as an orientation to the MBTR program at which time consents will be signed. Subjects will be randomly assigned to 2 groups of 32 participants, and at the completion of the 30-minute interview a research assistant will administer baseline psychometric assessments (see below for the list of measures used).

Primary Outcome Measures

• Tinnitus Handicap Inventory (THI) The THI is a self-report measure that can be used in a busy clinical practice to quantify the impact of tinnitus on daily living. The measure is brief, easy to administer and interpret, broad in scope, and psychometrically robust. Convergent validity was assessed using another measure of perceived tinnitus handicap (Tinnitus Handicap Questionnaire). Construct validity was assessed using the Beck Depression Inventory, Modified Somatic Perception Questionnaire, symptom rating scales (annoyance, sleep disruption, depression, and concentration), and perceived tinnitus pitch and loudness judgments. The THI is comprised of 25-item items grouped into functional, emotional, and catastrophic subscales. The total scales yield excellent internal consistency reliability (Cronbach's alpha=.93).

Secondary Outcome Measures

* Tinnitus Visual Analogue Scale (TVAS) Tinnitus Visual Analogue Scale (VAS) is a collection of straight lines 100mm in length anchored at the end with extremes (e.g., not bothersome, extremely bothersome) of the tinnitus sensation, feeling or response. The strength of this method lies in the compellation of several measurements (e.g., weekly average of tinnitus annoyance). This method of measuring distress has been recommended for use in research (Axelsson, Coles, Erlandsson, Meikle, & Vernon, 1993).
* Hospital Anxiety and Depression Scale (HADS) The HADS (Zigmond & Snaith, 1983) was chosen as a measure of self-reported depression and anxiety. As compared to the Beck Depression Inventory and State Trait Anxiety Inventory, the HADS is a 14 item questionnaire and does not tend to overburden or exhaust patients regarding filling out measures. The HADS is a more discrete measure that controls for complaints better explained by the somatic problem than does the BDI or STAI (Hermann, 1997).
* The Symptom Checklist-90-Revised (SCL-90-R) The Symptom Checklist-90-Revised (SCL-90-R) will be used to assess psychological distress (Derogatis 1983). SCL-90-R is a 90-item questionnaire measuring psychological distress over the past week. Reliability and validity of the measure is found to be high. The Global Severity Index (GSI) is used as a measure of overall psychological distress. The SCL-90-R has been used in several previous MBSR studies to measure psychological status (Kabat-Zinn, et al. 1992; Kabat-Zinn, et al. 1985; Kabat-Zinn, et al.1987; Kaplan, et al. 1993; Miller, et al. 1995; Majumdar, et al. 2002).
* Five Facet Mindfulness Questionnaire (FFMQ) Five-Facet Mindfulness Questionnaire (FFMQ; R. A. Baer, Smith, Hopkins, Krietemeyer, & Toney, 2006), is a 39-item inventory assessing five facets of mindfulness.

The FFMQ has been shown to have strong psychometric characteristics, including adequate to good internal consistencies for all facets and significant correlations in predicted directions with a variety of other constructs (R. A. Baer et al., 2006, 2008).

Description of MBTR Course The Mindfulness Based Tinnitus Reduction (MBTR) program is an 8-week course held one evening per week for 2 ½ hours. Participants will also complete a day-long Sunday retreat between the 6th and 7th sessions.

Modeled after the original Mindfulness Based Stress Reduction (MBSR) program developed by Jon Kabat-Zinn, PhD at the University of Massachusetts Medical Center, the MBTR course will introduce participants to mindfulness practice in the form of sitting meditation, body awareness and mindful movement, and informal mindfulness practices of daily life (e.g., eating, communicating, working, coping). Meditation will be introduced in four formats: sitting meditation using the breath as an anchor of attention, sitting meditation characterized by a state of open awareness, progressive body relaxation, and contemplative walking. Participants will be asked to practice at home for 30 minutes 6 days per week between sessions, aided by an audio CD. The two MBSR trained co-investigators will co-lead the classes. Participants will be provided with a copy of Full Catastrophe Living by Jon Kabat-Zinn, PhD. Intervention participants will be asked to document the number of minutes spent daily on each practice at home during their participation in the 8-week program.

MBTR Course Outline

The course in Mindfulness-Based Tinnitus Reduction (MBTR) takes place over eight weeks. Classes are approximately 2-1/2 hours long and are held in the evening once a week. Each class consists of guided meditations, gentle movement exercises, lecture, and group discussion as mindfulness relates to their experience with tinnitus. The course includes an all-day session on a Sunday between the sixth and seventh week. Between classes, subjects will enhance their participation through working with meditation CDs, homework assignments, and readings from the course materials and textbook. The in-class curriculum includes the following components:

* Week 1: Introduction to Program ° Foundations of Mindfulness ° More right with you than wrong ° Introduction to Body Scan meditation ° Tinnitus Discussion
* Week 2: Patience ° Working with perceptions °The Wandering Mind ° The STOP exercise
* Week 3: Non-Striving ° Introduction to Awareness of Breathing Meditation ° Mindful Yoga
* ° Attention vs. Disattention ° Tinnitus Discussion
* Week 4: Non-Judging ° Responding vs. Reacting ° Seeing Our Patterns ° Sitting Meditation
* ° Standing Yoga ° Research on Stress & Stress Hardiness ° Tinnitus Discussion
* Week 5: Acknowledgment ° Group Reflections on Halfway Point ° Small & Large Groups ° Sitting Meditation ° Qi Gong ° Tinnitus Discussion
* Week 6: Letting it Be ° Skillful Communication ° Avoiding Difficulty vs. Entering and Blending° Loving-kindness Meditation ° Walking Meditation ° Tinnitus Discussion

Daylong Session (see outline below)

* Week 7: Sitting Meditation ° Mindful Movement ° Trust & Self-Reliance ° Learning How to Practice on One's Own ° Mindfulness in Everyday Life ° Tinnitus Discussion
* Week 8: Sitting Meditation ° Mindful Movement ° The Class Never Ends: Practice for the rest of Your Life ° Course Review & Group Reflection

Mindfulness-Based Tinnitus Reduction Daylong Outline

The Mindfulness-Based Tinnitus Reduction Daylong (9:30am to 4:30pm between the 6th and 7th weeks) is part of the course and consists of a day of lead meditations, gentle movement exercises, and group sharing. A typical schedule is as follows:

9:30: Introductions 10:00: Awareness of Breathing 10:15: Yoga 10:30: Body Scan Meditation 11:15: Walking Meditation 11:45: Sitting Meditation 12:15: Lunch & Rest 1:30: Yoga 2:00: Sitting Meditation 2:30: Walking Meditation 2:45: Sitting Meditation 3:10: Walking Meditation 3:25: Lovingkindness Meditation 3:45: Group Discussion (Check Out) 4:30: Farewell

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* English speaking
* Duration of subjective chronic tinnitus > 6 months
* Moderate to strong tinnitus annoyance (Minimum THI score of > 28 )

Exclusion Criteria:

* Age < 18
* Non-English speaking
* > Moderate Hearing Loss
* Duration of chronic subjective tinnitus < 6 months
* Treatable tinnitus
* Severe depression and/or anxiety
* Recent (within 3-month) history of alcohol or drug abuse or dependence other than tobacco or caffeine
* No recent (within 3 months) start of new tinnitus treatment
* THI score < 28
* No previous psychological treatment for their tinnitus.
* History of traumatic brain injury (TBI) with loss of consciousness (LOC)
* History of psychotic disorders or dementia
* Currently undergoing litigation or legal matters related to auditory disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in Tinnitus Handicap Inventory (THI) | Baseline, Post-intervention (within 2 weeks after completion of 8-week intervention)
  The THI is a self-report measure that can be used in a busy clinical practice to quantify the impact of tinnitus on daily living. The measure is brief, easy to administer and interpret, broad in scope, and psychometrically robust. Convergent validity was assessed using another measure of perceived tinnitus handicap (Tinnitus Handicap Questionnaire). Construct validity was assessed using the Beck Depression Inventory, Modified Somatic Perception Questionnaire, symptom rating scales (annoyance, sleep disruption, depression, and concentration), and perceived tinnitus pitch and loudness judgments. Pre-assessment measures were individually administered to participants at the UCSF Audiology Clinic immediately after consents were signed, no earlier than 2 weeks prior to the start of the intervention. Post-assessment measures were filled out at home and mailed back to the Clinic by participants no more than 2 weeks after the intervention's completion.

SECONDARY OUTCOMES:
Change in Symptom Checklist-90- Revised | Baseline, Post-intervention (within 2 weeks after completion of 8-week intervention)
  Pre-assessment measures were individually administered to participants at the UCSF Audiology Clinic immediately after consents were signed, no earlier than 2 weeks prior to the start of the intervention. Post-assessment measures were filled out at home and mailed back to the Clinic by participants no more than 2 weeks after the intervention's completion.
Change in Five-Factor Mindfulness Questionnaire (FFMQ) | Baseline, Post-intervention (within 2 weeks after completion of 8-week intervention)
  Pre-assessment measures were individually administered to participants at the UCSF Audiology Clinic immediately after consents were signed, no earlier than 2 weeks prior to the start of the intervention. Post-assessment measures were filled out at home and mailed back to the Clinic by participants no more than 2 weeks after the intervention's completion.
Change in Hamilton Anxiety & Depression Scale (HADS) | Baseline, Post-intervention (within 2 weeks after completion of 8-week intervention)
  Pre-assessment measures were individually administered to participants at the UCSF Audiology Clinic immediately after consents were signed, no earlier than 2 weeks prior to the start of the intervention. Post-assessment measures were filled out at home and mailed back to the Clinic by participants no more than 2 weeks after the intervention's completion.
Change in Tinnitus Visual Analogue Scale (VAS) | Baseline, Post-intervention (within 2 weeks after completion of 8 week intervention)
  Tinnitus Visual Analogue Scale (VAS) is a collection of straight lines 100mm in length anchored at the end with extremes (e.g., no tinnitus distress, extreme tinnitus distress) of the tinnitus sensation, feeling or response. This means of measuring distress has been suggested for use in research (Axelsson, Coles, Erlandsson, Meikle, & Vernon, 1993). Pre-assessment measures were individually administered to participants at the UCSF Audiology Clinic immediately after consents were signed, no earlier than 2 weeks prior to the start of the intervention. Post-assessment measures were filled out at home and mailed back to the Clinic by participants no more than 2 weeks after the intervention's completion.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Gans, PsyD, Study Director — Clinical Psychologist
Locations (2):
- United States (2):
  - UCSF Audiology Clinic, San Francisco, California
  - UCSF, San Francisco, California

REFERENCES:
- [Background] Andersson G. Psychological aspects of tinnitus and the application of cognitive-behavioral therapy. Clin Psychol Rev. 2002 Sep;22(7):977-90. doi: 10.1016/s0272-7358(01)00124-6. PMID 12238249
- [Background] Grossman P, Tiefenthaler-Gilmer U, Raysz A, Kesper U. Mindfulness training as an intervention for fibromyalgia: evidence of postintervention and 3-year follow-up benefits in well-being. Psychother Psychosom. 2007;76(4):226-33. doi: 10.1159/000101501. PMID 17570961
- [Background] Henry, J. L., & Wilson, P. H. (2001). The psychological management of chronic tinnitus. Needham Heights, MA: Allyn & Bacon.
- [Background] Kabat-Zinn J, Massion AO, Kristeller J, Peterson LG, Fletcher KE, Pbert L, Lenderking WR, Santorelli SF. Effectiveness of a meditation-based stress reduction program in the treatment of anxiety disorders. Am J Psychiatry. 1992 Jul;149(7):936-43. doi: 10.1176/ajp.149.7.936. PMID 1609875
- [Background] Kabat-Zinn J, Lipworth L, Burney R. The clinical use of mindfulness meditation for the self-regulation of chronic pain. J Behav Med. 1985 Jun;8(2):163-90. doi: 10.1007/BF00845519. PMID 3897551
- [Background] Kabat-Zinn J, Wheeler E, Light T, Skillings A, Scharf MJ, Cropley TG, Hosmer D, Bernhard JD. Influence of a mindfulness meditation-based stress reduction intervention on rates of skin clearing in patients with moderate to severe psoriasis undergoing phototherapy (UVB) and photochemotherapy (PUVA). Psychosom Med. 1998 Sep-Oct;60(5):625-32. doi: 10.1097/00006842-199809000-00020. PMID 9773769
- [Background] Mason O, Hargreaves I. A qualitative study of mindfulness-based cognitive therapy for depression. Br J Med Psychol. 2001 Jun;74 Part 2:197-212. PMID 11802836
- [Background] Moller AR. Similarities between severe tinnitus and chronic pain. J Am Acad Audiol. 2000 Mar;11(3):115-24. PMID 10755808
- [Background] Pradhan EK, Baumgarten M, Langenberg P, Handwerger B, Gilpin AK, Magyari T, Hochberg MC, Berman BM. Effect of Mindfulness-Based Stress Reduction in rheumatoid arthritis patients. Arthritis Rheum. 2007 Oct 15;57(7):1134-42. doi: 10.1002/art.23010. PMID 17907231
- [Background] Sadlier M, Stephens SD, Kennedy V. Tinnitus rehabilitation: a mindfulness meditation cognitive behavioural therapy approach. J Laryngol Otol. 2008 Jan;122(1):31-7. doi: 10.1017/S0022215107007438. Epub 2007 Apr 23. PMID 17451612
- [Background] Speca, M., Carlson, L. E., Mackenzie, M. J., & Angen, M. (2006). Mindfulness-based stress reduction (MBSR) as an intervention for cancer patients. In R. A. Baer (Ed.), Mindfulness-based treatment approaches: Clinician's guide to evidence base and applications (pp. 239-261). San Diego, CA: Elsevier Academic Press.
- [Background] Surawy C, Roberts J, Silver A. (2005). The effect of mindfulness training on mood and measures of fatigue, activity, and quality of life in patients with chronic fatigue syndrome on a hospital waiting list: a series of exploratory studies. Behavioural and Cognitive Psychotherapy; 33:103-09
- [Background] Sweetow RW. Cognitive aspects of tinnitus patient management. Ear Hear. 1986 Dec;7(6):390-6. doi: 10.1097/00003446-198612000-00008. PMID 3792682
- [Background] Tonndorf J. The analogy between tinnitus and pain: a suggestion for a physiological basis of chronic tinnitus. Hear Res. 1987;28(2-3):271-5. doi: 10.1016/0378-5955(87)90054-2. PMID 2820913
- [Background] Williams, M., Teasdale, J., Zindel, S., Kabbat-Zinn, J.. (2007). The mindful way through depression. NY: The Guilford Press.